CLINICAL TRIAL: NCT05165836
Title: Role of Dexmedetomidine as Adjuvant With Bupivacaine in Ultrasound-Guided Erector Spinae Plane Block for Postoperative Analgesia After Shoulder Arthroscopy: A Randomized Controlled Study
Brief Title: Dexmedetomidine as Adjuvant in Erector Spinae Plane Block After Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKSU 40-11-21
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Arthroscopy; Erector Spinae Plane Block; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane block without Dexmedetomidine group (Placebo Comparator): Patients received Ultrasound-guided Erector Spinae Plane block at T2 using 19 ml of bupivacaine 0.25% + 1 mL saline
  Interventions: Procedure: Erector Spinae Plane block without Dexmedetomidine group
- Erector Spinae Plane block with Dexmedetomidine group (Experimental): Patients received Ultrasound-guided Erector Spinae Plane block at T2 using 19 ml of bupivacaine 0.25% + 1 mL dexmedetomidine 0.5 µg/kg
  Interventions: Procedure: Erector Spinae Plane block with Dexmedetomidine group

INTERVENTIONS:
Procedure: Erector Spinae Plane block without Dexmedetomidine group — Block will be performed with an ultrasound machine (Philips CX50 Extreme edition). A 2-5 MH2 curved probe will be positioned transversely to visualize the lateral tip of thoracic vertebrae2 transverse Process. Before surgery with patients in sitting position, the transducer will be positioned longitudinally 3 cm lateral to the thoracic vertebrae2 spinous process. The trapezius, rhomboid major, and erector spinae muscles will be revealed superficial to the shadow of the hyperechoic transverse process. Then, 3ml lidocaine 2% will be used to anesthetize the skin. Using a 20-gauge block needle put in-plane in a cephalad-to-caudad orientation to position the tip into the fascial plane on the deep (anterior) side of the erector spinae muscle, 19 ml of bupivacaine 0.25% + 1 mL saline will be injected. The needle tip's placement will be confirmed by observable fluid spread lifting the erector spinae muscle away from the transverse process's bony shadow.
  Arms: Erector Spinae Plane block without Dexmedetomidine group
Procedure: Erector Spinae Plane block with Dexmedetomidine group — Block will be performed with an ultrasound machine (Philips CX50 Extreme edition). A 2-5 MH2 curved probe will be positioned transversely to visualize the lateral tip of thoracic vertebrae2 transverse Process. Before surgery with patients in sitting position, the transducer will be positioned longitudinally 3 cm lateral to the thoracic vertebrae2 spinous process. The trapezius, rhomboid major, and erector spinae muscles will be revealed superficial to the shadow of the hyperechoic transverse process. Then, 3ml lidocaine 2% will be used to anesthetize the skin. Using a 20-gauge block needle put in-plane in a cephalad-to-caudad orientation to position the tip into the fascial plane on the deep (anterior) side of the erector spinae muscle, 19 ml of bupivacaine 0.25% + 1 mL dexmedetomidine 0.5 µg/kg will be injected. The needle tip's placement will be confirmed by observable fluid spread lifting the erector spinae muscle away from the transverse process's bony shadow.
  Arms: Erector Spinae Plane block with Dexmedetomidine group

SUMMARY:
The aim of this study is to evaluate the effect of adding dexmedetomidine as an adjuvant to bupivacaine in ultrasound (US) guided erector spinae plane block (ESPB) for managing acute postoperative pain in patients undergoing shoulder arthroscopy.

DETAILED DESCRIPTION:
Shoulder arthroscopy is a common procedure done is orthopedics for many surgical indications as rotator cuff tears, stiffness and instability. This procedure has a well - documented postoperative pain. To improve the outcome after surgery, effective pain control is needed.

There are many postoperative pain management modalities after shoulder arthroscopy including non-steroidal anti-inflammatory drugs, intraarticular injection, regional nerve blocks, patient controlled analgesia and cryotherapy.

The erector spinae plane block (ESPB) is one of the emerging regional techniques for managing postoperative pain. ESPB has been used successfully in many surgeries such as mastectomy, thoracotomies , percutaneous nephrolithotomies, lumbar fusions, hernia repair, cesarean delivery and even in total hip arthroplasty .

ESPB has been successfully used to treat chronic shoulder pain, and the local anesthetic spread was reported to reach the level of C3 when it was performed at T2.

Dexmedetomidine is a very selective α2 adrenoceptor agonist that is tenfold more selective than clonidine. It is a highly flexible medication in anesthetic practice, finding use in an expanding range of clinical circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Both genders and BMI < 40 kg/m2
* American Society of Anesthesiologists (ASA) physical status I-II
* Patients who are posted for elective shoulder arthroscopy

Exclusion Criteria:

* Known allergy to local anesthetics
* Allergy to all opioid medications
* Diagnostic shoulder arthroscopic procedures,
* Patients with chronic opioid use and coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The total rescue morphine (mg) consumption in the first 24 post-operative hours. | 24 hours postoperative
  Rescue analgesia in the form of 3 mg IV morphine (mg) will be given if the numeric rating scale (NRS) score is ≥ 4 repeated with 10 minutes lockout interval till the numeric rating scale (NRS) score becomes less than 3

SECONDARY OUTCOMES:
Post-operative pain score | 24 hours Postoperative
  After extubation, patients will be evaluated for pain using a numeric rating scale (NRS) score at 0,3,6,12,24 h for pain that ranged from (0 = no pain) to (10 = the worst imaginable pain). If the score is ≥ 4, rescue analgesia will be given in the form of fentanyl in a dose of 0.5µg/kg by iv route.
Time to first request of rescue analgesia | 24 hours Postoperative
  Time to the first rescue analgesic request (min) will be also recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El-Sheikh University Hospitals, Kafr ElSheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The supporting data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study

REFERENCES:
- [Derived] Hamed MA, Fargaly OS, Abdelghaffar RA, Moussa MA, Algyar MF. The role of dexmedetomidine as an adjuvant for high-thoracic erector spinae plane block for analgesia in shoulder arthroscopy; a randomized controlled study. BMC Anesthesiol. 2023 Feb 15;23(1):53. doi: 10.1186/s12871-023-02014-2. PMID 36793000